CLINICAL TRIAL: NCT06321523
Title: Clinical Benefit of Tafamidis 61mg for Transthyretin Amyloid Cardiomyopathy (ATTR-CM) Patients in Korean Population in the Real-world Setting, Multicenter, Non-interventional Study
Brief Title: A Study to Learn About the Study Medicine Called Tafamidis 61mg in People Diagnosed With Transthyretin Amyloid Cardiomyopathy (ATTR-CM)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B3461122; NCT06321523 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Transthyretin Amyloid Cardiomyopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ATTR-CM patients in Korea: transthyretin amyloid cardiomyopathy (ATTR-CM) patients in Korea
  Interventions: Drug: Tafamidis 61 milligrams

INTERVENTIONS:
Drug: Tafamidis 61 milligrams — Tafamidis 61mg as provided in real-world practice

SUMMARY:
The purpose of this clinical trial is to learn about the effects of the study medicine (called Tafamidis 61milligrams (mg)) for the potential treatment of Transthyretin amyloid cardiomyopathy (ATTR-CM).

This study is seeking participants who were prescribed Tafamidis 61mg after being diagnosed with ATTR-CM and have taken Tafamidis 61mg at least once.

We will examine the experiences of people receiving the study medicine. This will help us determine if the study medicine is safe and effective.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥19 years
* Patients diagnosed with ATTR-CM (ATTRwt and ATTRv) with tissue biopsy or nuclear scintigraphy
* Patients who was prescribed Tafamidis 61mg after being diagnosed with ATTR-CM and have taken Tafamidis 61mg at least once.

Exclusion Criteria:

* Presence of other amyloidosis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (more than 19 aged) who were prescribed Tafamidis 61mg after being diagnosed with ATTR-CM and have takne Tafamidis 61mg at least once.
  Participants will be enrolled through medical chart review from tertiary medical centers in Korea.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2025-10-13 (Actual); Study Completion 2025-10-13 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Change From Baseline in New York Heart Association (NYHA) Classification | baseline and 6, 12, 18, and 24 months after taking Tafamidis 61mg
Change from baseline in six-minute walk test | baseline and 6, 12, 18, and 24 months after taking Tafamidis 61mg
Change From Baseline in Kansas City Cardiomyopathy Questionnaire Overall Score (KCCQ-OS) | baseline and 6, 12, 18, and 24 months after taking Tafamidis 61mg
Change From Baseline in N-Terminal Prohormone Brain Natriuretic Peptide (NT-proBNP) Concentration | baseline and 6, 12, 18, and 24 months after taking Tafamidis 61mg
Change From Baseline in Troponin I and Troponin T | baseline and 6, 12, 18, and 24 months after taking Tafamidis 61mg
number of participants with Any Heart Block | baseline and 6, 12, 18, and 24 months after taking Tafamidis 61mg
number of participants with Atrioventricular (AV) block | baseline and 6, 12, 18, and 24 months after taking Tafamidis 61mg
Change From Baseline in Left Ventricular Ejection Fraction | baseline and 6, 12, 18, and 24 months after taking Tafamidis 61mg
Change From a Baseline in Diastolic function grades | baseline and 6, 12, 18, and 24 months after taking Tafamidis 61mg
Change from Baseline in Left Ventricular Wall Thickness | baseline and 6, 12, 18, and 24 months after taking Tafamidis 61mg
Change From Baseline in Global Longitudinal Strain scores | baseline and 6, 12, 18, and 24 months after taking Tafamidis 61mg

SECONDARY OUTCOMES:
Frequency of cardiovascular hospitalizations | Up to 24 months
Frequency of death due to any cause | Up to 24 months
  This includes participants who discontinue for transplantation (heart transplantation and combined heart and liver transplantation) or for implantation of a cardiac mechanical assist device.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- South Korea (4):
  - Severance Hopital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - Pusan National University Hospital, Busan
  - Gangnam Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B3461122